CLINICAL TRIAL: NCT03405792
Title: Phase 2, Single Arm, Historically Controlled Study Testing The Safety and Efficacy of Adjuvant Temozolomide Plus TTFields (Optune®) Plus Pembrolizumab in Patients With Newly Diagnosed Glioblastoma (2-THE-TOP)
Brief Title: Study Testing The Safety and Efficacy of Adjuvant Temozolomide Plus TTFields (Optune®) Plus Pembrolizumab in Patients With Newly Diagnosed Glioblastoma (2-THE-TOP)
Acronym: 2-THE-TOP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702270; OCR16397 (Other: University of Florida)
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Glioblastoma, WHO Grade IV
Keywords: Tumor Treating Electric Fields (TTFields)
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optune System combined with Temozolomide (TMZ) + Pembrolizumab (Experimental): Patients with newly-diagnosed GBM who undergo maximal safe resection (biopsy alone is eligible) followed by chemoradiation consisting of concomitant TMZ daily and radiation therapy (RT) with minimal RT will be eligible for this trial. Four to six weeks after finishing chemoradiation, patients will start monthly cycles of adjuvant TMZ. Treatment with Optune will start at approximately the same time as the first cycle of adjuvant TMZ and continue until second disease progression or a maximum of 2 years. Within one week after starting Cycle 2 of adjuvant TMZ and Optune therapy, patients will begin open-label treatment with pembrolizumab every 3 weeks until first disease progression or unacceptable toxicities or 2 years, whichever comes first.
  Interventions: Drug: Temozolomide (TMZ); Device: Optune System; Drug: Pembrolizumab
- Historical Control (Other): Historical control of patients treated with Optune System combined with Temozolomide alone from the EF-14 study will be compared with the Optune System combined with Temozolomide (TMZ) + pembrolizumab
  Interventions: Drug: Temozolomide (TMZ); Device: Optune System

INTERVENTIONS:
Drug: Temozolomide (TMZ) — Patients will begin treatment with adjuvant TMZ at least 4 weeks but no more than 6 weeks from last dose of concomitant temozolomide or radiation therapy (the latter of the two). A minimum of 6 and maximum of 12 cycles of adjuvant TMZ will be given depending on tolerability and toxicity.
Device: Optune System — Patients will undergo 24-months of planned treatment with Optune therapy.
  Other Names: NovoTTF Therapy
Drug: Pembrolizumab — Pembrolizumab will be given intravenously every 3 weeks beginning on Day 1 of Cycle 2 of adjuvant TMZ. Treatment with pembrolizumab every 3 weeks until first disease progression or unacceptable toxicities or 2 years, whichever comes first.
  Other Names: Keytruda
  Arms: Optune System combined with Temozolomide (TMZ) + Pembrolizumab

SUMMARY:
Glioblastoma multiforme (GBM) is the most common and deadliest primary malignant neoplasm of the central nervous system in adults. Despite an aggressive multimodality treatment approach including surgery, radiation therapy and chemotherapy, overall survival remains poor. Pembrolizumab has recently been approved in the United States for the treatment of patients with advanced and metastatic non-small cell lung cancer, recurrent or metastatic head and neck squamous cell carcinoma, locally advanced urothelial carcinoma, classical Hodgkin lymphoma, unresectable or metastatic melanoma

This study is being performed to determine whether the triple combination of pembrolizumab when added to TTFields (Optune®) and adjuvant temozolomide increases progression-free survival (PFS) in patients with newly diagnosed GBM as compared to historical control data.

DETAILED DESCRIPTION:
Patients with newly-diagnosed GBM who undergo maximal safe resection (biopsy alone is eligible) followed by standard chemoradiation will be eligible for this trial.

Four weeks after completing chemoradiation, patients will undergo baseline standard of care MRI. Four to six weeks after finishing chemoradiation, patients will start monthly cycles of adjuvant TMZ. A minimum of 6 and maximum of 12 cycles of adjuvant TMZ will be given. Treatment with Optune will start at approximately the same time as the first cycle of adjuvant TMZ and continue until second disease progression or a maximum of 2 years. Within one week after starting Cycle 2 of adjuvant TMZ and Optune therapy, patients will begin open-label treatment with pembrolizumab every 3 weeks until first disease progression or unacceptable toxicities or 2 years, whichever comes first.

At first progression, patients will be allowed to continue with Optune therapy combined with any other therapy, which may include pembrolizumab, per standard of care at the discretion of the treating physician. Surgical resection or biopsy of first recurrent tumor for confirmation of recurrence is allowed within the protocol.

All patients will be seen before Cycle 1 of TMZ, before cycle 2 of TMZ, before starting the second dose of pembrolizumab, and every 3 weeks before each subsequent pembrolizumab dose at an outpatient clinic until they complete all 12 cycles of adjuvant TMZ or discontinue TMZ due to toxicity or first progression.

Medical follow-up will continue for 30 days after treatment termination. After this visit, mortality will be assessed based on telephone interviews with the patients or the patients' caregivers every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of glioblastoma, WHO Grade IV (GBM variants are allowed; Lower grade gliomas that have been transformed to GBM will be considered newly diagnosed GBM if the lower-grade tumor was not previously treated, and the standard treatment for GBM including radiation and temozolomide is now planned).
* MGMT methylation status if available (indeterminate methylation status will be considered unmethylated).
* Karnofsky performance status (KPS) ≥70%.
* Patients must be at least 18 years of age.
* Received maximal safe resection (biopsy only allowed) and radiotherapy concomitant with temozolomide:

  1. Gliadel wafers placement at the time of surgical resection is allowed.
  2. Any additional treatment directed at GBM will be considered exclusionary.
  3. Minimum dose for concomitant radiotherapy is 40 Gy.
* Candidate for adjuvant high dose temozolomide and Optune therapy.
* Life expectancy of at least 3 months.
* Adequate bone marrow and organ function as defined below:

  1. ANC ≥ 1,500/mcL
  2. Platelets ≥ 100,000/mcL
  3. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L (transfusion is allowed)
  4. Serum creatinine ≤ 1.5 x IULN OR creatinine clearance by Cockcroft-Gault ≥ 60 mL/min for patients with serum creatinine > 1.5 x IULN
  5. Serum total bilirubin ≤ 1.5 x IULN OR direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
  6. AST (SGOT) and ALT (SGPT) ≤ 3 x IULN
* Participants of childbearing age must use effective contraception:

  * Women of childbearing potential (WOCBP) must be using a highly effective method of contraception to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Refer to Appendix D for guidance on highly effective contraceptive methods.
  * WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or oophorectomy) or who is not post-menopausal. Post-menopause is defined as:
  * Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
  * For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
  * Males with female partners of childbearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.
* Ability of the patient or their legally authorized representative (LAR) to understand and willingness to sign an IRB approved written informed consent document
* Steroid dose equivalent to dexamethasone dose of ≤ 4mg daily at the time of starting adjuvant treatment
* Optune and temozolomide treatment start date will be at least 4 weeks but not more than 6 weeks from the later of last dose of concomitant temozolomide or radiotherapy. Although Optune and temozolomide should be started simultaneously, it is not required as long as both are started within this time frame

Exclusion Criteria:

* Prior treatment with anti-angiogenic agents including bevacizumab.
* History of other malignancy that, in the primary oncologist's estimation, has a higher risk of recurrence or death than the study-related cancer at the time of study participation.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Progressive disease (according to RANO criteria). Advanced imaging is allowed to further investigate suspected pseudoprogression if deemed necessary.
* Actively participating in another clinical treatment trial intended to treat GBM.
* Multifocal gliomas defined as distinct tumors that do not have overlapping T2/FLAIR signal.
* Presence of leptomeningeal metastases.
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
* Tumor is entirely located in the infra-tentorial region.
* History of hypersensitivity reactions or allergies to hydrogels and/or compounds of similar chemical or biologic composition to Temozolomide and Pembrolizumab.
* Steroid dose equivalent to > 4 mg dexamethasone at the time of starting adjuvant therapy.
* History of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (with the exception of daily dexamethasone ≤ 4 mg).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Pregnant and/or breastfeeding. Patient must have a negative serum or urine pregnancy test within 72 hours of study entry.
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 24 weeks after the last dose of study drug.
* Known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected) infection.
* Known history of active TB (bacillus tuberculosis).
* Known history of HIV (HIV 1/2 antibodies).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen D, Le SB, Ghiaseddin AP, Manektalia H, Li M, O'Dell A, Rahman M, Tran DD. Efficacy and safety of adjuvant TTFields plus pembrolizumab and temozolomide in newly diagnosed glioblastoma: A phase 2 study. Med. 2025 Sep 12;6(9):100708. doi: 10.1016/j.medj.2025.100708. Epub 2025 Jun 4. PMID 40466642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in 2018 and lasted until July 2021. Patients with newly diagnosed GBM who completed standard of care radiation therapy together with concomitant TMZ were recruited. Neuro-oncologists identified subjects as part of routine clinical care. Patients with newly-diagnosed GBM who underwent maximal safe resection followed by chemoradiation consisting of concomitant TMZ 75mg/m2 daily and RT with minimal RT dose of 40gy were eligible for this trial.
Pre-assignment Details: Four to 6 weeks post- chemoradiation, patients began monthly cycles of adjuvant TMZ (minimum 6 and maximum 12 cycles of adjuvant TMZ) and treatment with Optune. Patients began treatment with pembrolizumab no sooner than 3 weeks after starting Optune therapy.
  Forty participants were consented. Nine were deemed ineligible. Five who were eligible to participate withdrew or were withdrawn because they did not start or discontinued Optune or did not receive pembrolizumab.
Groups:
- Historical Control: Historical control data of patients treated with Optune System combined with Temozolomide alone will be compared with the Optune System combined with Temozolomide (TMZ) + Pembrolizumab arm.
  Temozolomide (TMZ): Patients will begin treatment with adjuvant TMZ at least 4 weeks but no more than 6 weeks from last dose of concomitant temozolomide or radiation therapy (the latter of the two). A minimum of 6 and maximum of 12 cycles of adjuvant TMZ will be given depending on tolerability and toxicity.
  Optune System: Patients will undergo 24-months of planned treatment with Optune therapy.
Period: Overall Study
Arm/Group | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab | Historical Control
Started | 31 | 466
Completed | 26 | 466
Not Completed | 5 | 0
Not completed — o Did not start or discontinued TTF during cycle 1 of TMZ for personal reasons | 4 | 0
Not completed — o Did not receive pembrolizumab | 1 | 0

BASELINE CHARACTERISTICS:
Population: Thirty-one participants were eligible. Twenty-six participants were treated with the combination of optune, adjuvant temozolomide and pembrolizumab and counted toward the primary outcome measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab | Historical Control | Total
Number analyzed (Participants) | 31 | 466 | 497
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 377 | 399
  >=65 years | 9 | 89 | 98
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.5 [49.1 to 67] | 56 [19 to 83] | NA [NA to NA] — We do not have the distribution of ages for the historical control arm to determine the median for the total population.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 150 | 159
  Male | 22 | 316 | 338
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 18 | 19
  Not Hispanic or Latino | 30 | 447 | 477
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 27 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 416 | 444
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 19 | 19
Region of Enrollment [Number; unit: participants]
  United States | 31 | 221 | 252

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Between the Groups From Time of Enrollment
Description: Time from enrollment to progression or death or censoring, whichever occurs first. The study team will use the one-sample log-rank test to compare PFS in the triple combination arm relative to the historical control arm to determine whether the triple combination treatment increases PFS in newly diagnosed GBM patients when compared to TTFields+TMZ historical control patients from the EF-14 study. Evaluability for progression free survival required participants to receive adjuvant TMZ, Optune and at least 1 dose of pembrolizumab.
Time Frame: Assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab | Historical Control
Number analyzed (Participants) | 26 | 466
months | 11.79 [8.71 to 22.72] | 6.7 [6.1 to 8.1]
Statistical Analysis 1: Comparison: Optune System Combined With Temozolomide (TMZ) + Pembrolizumab; We will use one-sample log-rank test to compare PFS between the triple combination arm relative to the historical control arm; Test type: Other; We took a look at median survival time and CI of our population and we compared it to the median PFS and CI of the historical control descriptively. There is no yielded P value

2. Secondary Outcome: Number of Participants With Toxicities, Serious Adverse Events and/or Other Adverse Events Treated With Triple Combination Treatment
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting for grade 3 or higher. We will estimate proportions and 95% confidence intervals for patients in the triple combination arm who experience toxicities and other types of AEs and serious AEs.
Time Frame: Assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab
Number analyzed (Participants) | 26
Participants | 26
Statistical Analysis 1: Comparison: Optune System Combined With Temozolomide (TMZ) + Pembrolizumab; Test type: Other; Every participant (26/26; 100%) experienced an adverse event

3. Secondary Outcome: Overall Survival (OS)
Description: Time from enrollment to death or censoring, whichever occurs first. We will use the log-rank test to compare OS between the triple combination arm relative to the historical control arm.
Time Frame: Assessed up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Augmentation of TTFields-initiated Glioma-specific Immune Reaction by Pembrolizumab
Description: We will use mixed effect regression to assess changes in response variables related to glioma-specific immune reaction before, during, and after treatment with pembrolizumab.
Time Frame: Assessed up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the initiation of treatment with the adjuvant treatment with TMZ and the Optune device, and ended at least 30-days following last study treatment for up to 24 months. Twenty-eight participants met criteria for AE collection; two of those did not receive pembrolizumab.
Description: Adverse event (AE) data for historical controls was reported and presented by Stupp et al. 2017. 466 patients were randomized to treatment in the TMZ+TTFields arm (the comparator for this study); 10 didn't complete treatment. For all cause mortality, we used the intent to treat population (all patients randomized to receive the intended treatment regardless of whether they completed) which was 466. AEs/SAEs were monitored/assessed for the 456 participants who completed the intended treatment.
Groups:
- Historical Control Optune System Combined With Temozolomide (TMZ): Historical control of patients treated with Optune System combined with Temozolomide alone from the EF-14 study based on data published by Stupp et al, 2017.
Arm/Group | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab | Historical Control Optune System Combined With Temozolomide (TMZ)
All-Cause Mortality (participants affected / at risk) | 25/28 | 265/466
Serious Adverse Events (participants affected / at risk) | 18/28 | 0/456
Other Adverse Events (participants affected / at risk) | 28/28 | 218/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab (N=28) | Historical Control Optune System Combined With Temozolomide (TMZ) (N=456)
Edema, head and neck (Blood and lymphatic system disorders) | 1 | 0
Platelets, thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Allergy/Immunology (Immune system disorders) | 1 | 0
Infection (Infections and infestations) | 6 | 0
Confusion (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 2 | 0
Memory Impairment (Nervous system disorders) | 1 | 0
Neurology, other (Nervous system disorders) | 2 | 0
Pain, Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Bruising (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Intra-operative injury - Brain (Surgical and medical procedures) | 8 | 0
Intra-operative injury, Acute Kidney Injury (Surgical and medical procedures) | 1 | 0
Intra-operative injury, extremity-lower (Surgical and medical procedures) | 1 | 0
Intra-operative injury, muscle (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Generalized Edema (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Optune System Combined With Temozolomide (TMZ) + Pembrolizumab (N=28) | Historical Control Optune System Combined With Temozolomide (TMZ) (N=456)
Gastrointestinal Disorders (Gastrointestinal disorders) | 22 | 23
Blood and Bone Marrow (Blood and lymphatic system disorders) | 9 | 59
Infections (Infections and infestations) | 11 | 32
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 10 | 24
Metabolism (Metabolism and nutrition disorders) | 3 | 16
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 19 | 21
Nervous System Disorders (Nervous system disorders) | 21 | 109
Respiratory (Respiratory, thoracic and mediastinal disorders) | 8 | 24

LIMITATIONS AND CAVEATS:
Limitation 1: We do not have the distribution of ages for the historical control arm to determine the median for the total population.

Limitation 2: Adverse Events for historical controls were monitored/assessed/reported without regard to the specific Adverse Event Term therefore we are not reporting for the historical control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03405792/Prot_SAP_000.pdf